CLINICAL TRIAL: NCT02389140
Title: Blood Flow Within Active Myofascial Trigger Points Following Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14-1582; UL1TR001082 (NIH)
Record Dates: First submitted 2015-03-02; First posted 2015-03-17 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Myofascial Pain; Tension-type Headache
Keywords: Blood flow; Glucose; lactic acid
MeSH Terms: conditions — Tension-Type Headache | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trigger point treatment (Experimental): Trigger point release
  Interventions: Other: Trigger point release
- Ultrasound (Sham Comparator): Sham US at Trigger point
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Trigger point release — Trigger point therapy
  Arms: Trigger point treatment
Other: Ultrasound — sham ultrasound
  Arms: Ultrasound

SUMMARY:
The physiological response at the myofascial trigger point (MTrP) to massage is not known, yet would provide important objective evidence for a treatment effect and clarify the resolution process of a MTrP.

DETAILED DESCRIPTION:
The physiological response at the myofascial trigger point (MTrP) to massage is not known, yet would provide important objective evidence for a treatment effect and clarify the resolution process of a MTrP. The long-term goal is to understand how therapeutic intervention affects the physiology of the MTrP. The objective of the proposed research is to assess, in a placebo controlled trial, the effectiveness of trigger point release massage (also known as ischemic compression) on blood flow at an active MTrP. The central hypothesis is that the contraction nodule of an active MTrP is characterized by an ischemic state comprised of reduced blood flow and subsequent dysregulation in carbohydrate metabolism. The investigators hypothesize that trigger point release (TPR) can positively impact blood flow leading to a change in high energy carbohydrate tension. The present study has been formulated, in part, from a preliminary study conducted by the investigators, which supports reduced blood flow and physiological disruption at active MTrPs. The proposed research will provide a physiological basis for massage to corroborate subjective reports of reduced pain sensitivity, impart credibility to treatment techniques, and provide insight into a mechanism of action for healing the MTrP.

ELIGIBILITY:
Inclusion Criteria:

* Chronic or episodic tension-type headache
* active MTrP in upper trapezius
* age 21-49
* BMI between 18.5-24.9
* either gender
* any race or ethnicity

Exclusion Criteria:

* No or latent MTrP in the upper trapezius
* migraine 4+/month
* cluster headache
* fibromyalgia
* neurological disease (e.g. Alzheimer's disease, Parkinson's disease, muscular dystrophy, multiple sclerosis)
* cardiovascular disease (e.g. prior heart attack or stroke)
* diabetes
* pregnancy
* a bleeding disorder (Self-report of hemophilia, known lack/deficiency of clotting factors, or presently °taking anti-coagulants (e.g. warfarin, Coumadin))
* narcotic use
* currently receiving massage
* prior trigger point injection or needling therapies
* allergy to lidocaine-type anesthetics such as lidocaine and prilocaine

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Blood Flow as measured by microdialysis | 1 hr pre intervention and 1 hr post intervention

SECONDARY OUTCOMES:
Change in Glucose as measured by microdialysis | 1 hr pre intervention and 1 hr post intervention
Change in Lactate as measured by microdialysis | 1 hr pre intervention and 1 hr post intervention
Change in Pyruvate as measured by microdialysis | 1 hr pre intervention and 1 hr post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Albert Moraska, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Derived] Moraska AF, Hickner RC, Rzasa-Lynn R, Shah JP, Hebert JR, Kohrt WM. Increase in Lactate Without Change in Nutritive Blood Flow or Glucose at Active Trigger Points Following Massage: A Randomized Clinical Trial. Arch Phys Med Rehabil. 2018 Nov;99(11):2151-2159. doi: 10.1016/j.apmr.2018.06.030. Epub 2018 Aug 6. PMID 30092205